CLINICAL TRIAL: NCT02790892
Title: Creative Arts Diabetes Initiative: Group Art Therapy and Peer Support for Youth and Young Adults Transitioning From Pediatric to Adult Diabetes Care
Brief Title: Creative Arts Diabetes Initiative for Youth/Young Adults Transitioning to Adult Care
Acronym: CADI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HS19577 (H2016:119)
Record Dates: First submitted 2016-05-25; First posted 2016-06-06 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Coping Behavior; Emotional Distress; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: type 1 diabetes; type 2 diabetes; children; adolescents; young adults; youth; transition; art therapy; behavioral therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Art therapy - pre and post test measures (Other): 20 young adults aged 15-24 years with diabetes (10 with type 1 diabetes and 10 with type 2 diabetes) receiving 12 weeks of group art therapy. Participants serve as their own controls.
  Interventions: Behavioral: Art therapy - pre and post test measures

INTERVENTIONS:
Behavioral: Art therapy - pre and post test measures — 12 weeks of 90 minutes of art therapy with pre and post test measures to determine changes in social support and levels of diabetes distress

SUMMARY:
The Creative Arts Diabetes Initiative will offer facilitated art therapy with a group/peer-support environment to two groups of youth/young adults, one with type 1 diabetes, and one with type 2 diabetes. This environment intends to "meet youth where they are", promote universality, hope and self-understanding, has the potential to be therapeutic and allows youth to express and learn about themselves and each other while developing healthy coping skills and address their fears and concerns.

DETAILED DESCRIPTION:
The Creative Arts Diabetes Initiative will offer facilitated art therapy with a group/peer-support environment to two groups of youth/young adults, one with type 1 diabetes, and one with type 2 diabetes. This environment intends to "meet youth where they are", promote universality, hope and self-understanding, has the potential to be therapeutic and allows youth to express and learn about themselves and each other while developing healthy coping skills and address their fears and concerns.

As much of diabetes management is about meeting physical health goals - it is the vision of this study that offering additional support in the form of art therapy will have positive effects for bringing awareness and avenues for self-care to the other often neglected dimensions of patients' mental, emotional and spiritual health as part of a more holistic health process.

Engaging in art therapy has the potential to decrease diabetes related distress by giving youth a means and opportunity to identify, understand and express their feelings about having diabetes. Improved self-awareness and self-reflectiveness can help youth integrate their feelings and learn how this can motivate, influence and impact their behaviors and life choices.

Youth will have the opportunity for engaging in peer support, and to build relationships that are meaningful, thus increasing their sense of belonging and positively affect their level of self-confidence, purpose and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with either type 1 or type 2 diabetes, live within weekly travel distance to Winnipeg, Manitoba, receive their pediatric care at the Diabetes Education Resource for Children and Adolescents, or who are members of the Maestro Project

Exclusion Criteria:

* those who cannot give informed consent or who are not able to attend regular sessions due to travel distance

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Decrease diabetes related distress | 12 weeks
  Decrease diabetes related distress as measured by the Diabetes Attitudes Wishes and Needs Study (DAWN) Problem Areas in Diabetes Questionnaire (PAID).

SECONDARY OUTCOMES:
Increase social support | 12 weeks
  Increase emotional and social support for youth as measured by Measures of Support (MOS) Social Support Survey.
Increase emotional | 12 weeks
  Increase emotional and social support for youth as measured by Mental Health Continuum Short Form (MHC-SF)

CONTACTS AND LOCATIONS:
Overall Officials: Seth D Marks, MD,MSc,FRCPC, Principal Investigator — University of Manitoba, Pediatric Endocrinology
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: young adult diabetes transition support service — http://www.maestroproject.com